CLINICAL TRIAL: NCT04548245
Title: Markers of Executive Attention Development in Preschoolers
Acronym: MEDiATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01503-36
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-03

CONDITIONS: Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term
  Interventions: Device: EEG
- Preterm
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — EEG

SUMMARY:
This project aims to identify precursors of executive attention that can serve as early markers of ADD.

ELIGIBILITY:
Inclusion Criteria:

* Normal schooling
* Parental consent

Exclusion Criteria:

- Psychotropic drug

Ages: 48 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschool children born preterm vs term
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Amplitude in µV of EEG changes relative to baseline when expected stimulus is omitted in a tactile stimulation sequence | at 4 years old

CONTACTS AND LOCATIONS:
Locations (1):
- Comete U1075 Inserm Unicaen, Caen, France

IPD SHARING:
Plan to Share IPD: No